CLINICAL TRIAL: NCT01524640
Title: A Randomized, Double-blind, Controlled Trial to Evaluate the Safety and Immunogenicity of Killed Bivalent (o1 and o139) Whole-cell Based Oral Cholera Vaccine (Shanchol®) in Healthy Individuals in Ethiopia
Brief Title: Bridging Study for Killed Oral Cholera Vaccine in Ethiopia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: International Vaccine Institute (Other)
Collaborators: Armauer Hansen Research Institute, Ethiopia (Other); Ministry of Health, Ethiopia (Other Government); Shantha Biotechnics Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CR-WC-09
Record Dates: First submitted 2012-01-31; First posted 2012-02-02 (Estimated); Last update posted 2015-05-04 (Estimated); Status verified 2015-05

CONDITIONS: Vibrio Cholerae; Cholera
Keywords: oral cholera vaccine; safety and immunogenicity; bridging study; ethiopia
MeSH Terms: conditions — Cholera

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Killed oral cholera vaccine (Experimental): Killed Bivalent (O1 and O139) Whole cell oral cholera vaccine (Shanchol TM) Vaccine strain Reformulated version
  V. cholerae O1 Inaba El Tor strain Phil 6973 formalin killed 600 Elisa units (EU) of lipopolysaccharide (LPS) V. cholerae O1 Ogawa classical strain Cairo 50 heat killed 300 EU LPS V. cholerae O1 Ogawa classical strain Cairo 50 formalin killed 300 EU LPS V. cholerae O1 Inaba classical strain Cairo 48 heat killed 300 EU LPS V. cholerae O139 strain 4260B formalin killed 600 EU LPS
  Interventions: Biological: Killed Bivalent (O1 and O139) whole cell oral cholera vaccine
- Placebo (Placebo Comparator): Non biologic placebo
  Ingredients Per 1.5 ml dose
  1. Starch 60mg
  2. Red color[1mg/ml] 10 µl
  3. Yellow color [1mg/ml] 5 µl
  4. Xanthum Gum (1% solution) 300 µl
  5. Water for Injection Upto 1.5 ml
  All the above ingredients are of pharmaceutical grade.
  Non-biological placebo of above composition has been used in 2010 for "Randomized, double-blind, placebo controlled trial to evaluate the safety and immunogenicity of orally administered, killed, bivalent whole-cell , cholera vaccine, Shanchol in Bangladeshi Adults and Children". This study involving 330 subjects was carried out at International Center for Diarrheal Disease Research Bangladesh (ICDDR,B) located in Dhaka, Bangladesh with Dr. Firdausi Qadri as Principal Investigator (NCT01042951). There were no safety concerns associated with this placebo in this study and the report of this study has been submitted to the National Regulators in Bangladesh and the World Health Organization.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Killed Bivalent (O1 and O139) whole cell oral cholera vaccine — 1.5 ml single dose oral administration on day 0 and day 14
  Other Names: Shanchol TM
  Arms: Killed oral cholera vaccine
Biological: Placebo — 1.5 ml oral administration on day 0 and day 14
  Other Names: Non biologic placebo
  Arms: Placebo

SUMMARY:
This is a randomized, double blind, placebo controlled trial to confirm the safety and determine the immune response of the killed oral cholera vaccine in healthy adults and children in Ethiopia.

DETAILED DESCRIPTION:
This study serves as a bridging trial to evaluate the safety and immunogenicity of a two dose regimen of the WC-OCV (Shanchol®) in Ethiopian population. In order to assess whether the bivalent killed oral cholera vaccine may be used safely among those who are most at risk for cholera, we need to determine the safety and immunogenicity of the killed oral cholera vaccine. The vaccine was evaluated in a large number of human subjects in India Vietnam, and Bangladesh, in which it has demonstrated safety, immunogenicity, and clinical protective efficacy. Though we do not expect the vaccine to act differently in the Ethiopian population, we aim to confirm our presumptive understanding that two doses of WC-OCV is safe and immunogenic in healthy volunteers at one year and above (exclusive of pregnant women). Findings from this study can pave the way for the possible use of the killed whole cell oral cholera vaccine in both endemic and outbreak settings at a larger scale.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female adults aged 18 years and above; and children aged 1 -17 years who is available for follow-up visits and specimen collection.

   * The subject should be able to continue in the study for the next 4 weeks
   * The subject (or parent/guardian) should be willing to provide 3 blood samples
2. For females of reproductive age, non-pregnant (as determined by urine pregnancy test).
3. Written informed consent obtained from the subjects or their parents/guardians, and written assent obtained from children aged 12 - 17 years.
4. Healthy subjects as determined by:

   * Medical history
   * Physical examination
   * Clinical judgment of the investigator

Exclusion Criteria:

1. Ongoing chronic recurring illness which may cause systemic symptoms as judged by the investigating physician.
2. Ongoing acute illness.
3. For females of reproductive age: Pregnancy (or females planning to become pregnant during the study period; as determined by verbal screening)
4. Immunocompromising condition or on chronic systemic steroid therapy
5. Diarrhea (3 or more loose/more watery stools within a 24-hour period) within 6 weeks prior to enrollment
6. Intake of any anti-diarrhea medicine in the past week
7. Abdominal pain or cramps, loss of appetite, nausea, or vomiting in the past 24 hours
8. Temperature ≥38ºC (oral or axillary) warrants deferral of the vaccination pending recovery of the subject
9. Previous hypersensitivity to formaldehyde.
10. Receipt of immunoglobulin or any blood product during the past 3 months
11. Receipt of oral cholera vaccine in the past three years
12. Any potential subject currently participating or who will participate within the next six months in another clinical trial
13. Positive screening urine pregnancy test for females greater than 12 years of age

Min Age: 1 Year | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2012-12; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects given investigational product with adverse events. | 6 months
  1. Immediate reactions within 30 minutes after each dose
  2. Serious Adverse Events occurring 14 days following each dose
  3. Reactogenicity: Headache, vomiting, nausea, abdominal pain/cramps, diarrhea, fever, loss of appetite within three days
  i. Diarrhea is defined as having 3 or more loose/watery stools within a 24 hour period.
  ii. Fever is defined as having an oral or axillary temperature of ≥ 38oC
Proportion of subjects exhibiting 4-fold or greater rises in titers of serum vibriocidal antibodies, relative to baseline, 14 days after second dose. | 6 months

SECONDARY OUTCOMES:
Proportion of subjects exhibiting 4-fold or greater rises in titers of serum vibriocidal antibodies, relative to baseline, 14 days after the first dose. | 6 months
Geometric mean serum vibriocidal titers at baseline, 14 days after each dose of the investigational product. | 6 months
Severe adverse event within 28 days following each dose of investigational product. | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Armauer Hansen Research Institute, Addis Ababa, Oromiya, Ethiopia

REFERENCES:
- [Derived] Desai SN, Akalu Z, Teshome S, Teferi M, Yamuah L, Kim DR, Yang JS, Hussein J, Park JY, Jang MS, Mesganaw C, Taye H, Beyene D, Bedru A, Singh AP, Wierzba TF, Aseffa A. A Randomized, Placebo-Controlled Trial Evaluating Safety and Immunogenicity of the Killed, Bivalent, Whole-Cell Oral Cholera Vaccine in Ethiopia. Am J Trop Med Hyg. 2015 Sep;93(3):527-533. doi: 10.4269/ajtmh.14-0683. Epub 2015 Jun 15. PMID 26078323